CLINICAL TRIAL: NCT04413019
Title: Planned Domiciliary Versus Hospital Care for Women With Preterm Prelabor Rupture of the Membranes (PPROM)
Brief Title: Domiciliary Versus Hospital Management of PPROM
Acronym: PPROM
Status: Completed | Type: Observational
Sponsor: Ahmed Mohammed Selim (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohammed Selim, ASelim, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: PPROM
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group (D): Planned domiciliary care.: Patients within this group will be counseled for home care with self-monitoring for any symptoms suggestive of preterm labor, maternal or fetal distress.
  Interventions: Other: Clinical follow up
- Group (H): Planned hospital care.: Patients within this group will be admitted at hospital for close monitoring of maternal & fetal wellbeing & finally the neonatal outcome
  Interventions: Other: Clinical follow up

INTERVENTIONS:
Other: Clinical follow up — Patients recruited in this study commenced antibiotic treatment according to the recent guidelines :
  * Erythromycin 250 mg 4 times daily for 10 days following the diagnosis of PPROM, or until the women is established labor (whichever sooner)
  * Penicillin may be used in patients who can't tolerate erythromycin
  * In cases of penicillin allergy: Cefazolin 1 g intravenously every 8 hours for 48 hours, followed by cephalexin 500 mg orally four times daily for five days. These drugs provide coverage for both GBS and Escherichia coli, the two major causes of neonatal infection.

SUMMARY:
This study is designed to compare efficacy & safety of planned domiciliary versus hospital care for women with preterm prelabor rupture of the membranes (PPROM) on fetal, neonatal and maternal outcome.

DETAILED DESCRIPTION:
Background: PPROM is encountered in 2.0% to 3.5% of pregnancies. Domiciliary care management is developing more and more in obstetrics, with psychological benefits for patients as well as other financial benefits. Reliable discharge criteria have been mentioned by few studies for patients with PPROM. Studies had shown that domiciliary care management in a context of PPROM did not modify perinatal morbidity and mortality, and allows a prolongation of the latency period. However, eligibility criteria for domiciliary care management were heterogeneous

Aim of The Work: The aim of this study is to compare efficacy & safety of planned domiciliary versus hospital care for women with preterm prelabor rupture of the membranes (PPROM) on fetal, neonatal and maternal outcome.

Patients & Methods: The current trial was conducted at Ain Shams University Maternity Hospital. A total of 3662 pregnant women were recruited from the outpatient clinic & emergency room and included in the study. Then, they were randomized into two groups; group (D) was counseled for home care management, while group (H) was hospitalized. Take-home baby was assessed as a primary outcome and other maternal, fetal & neonatal complications were recorded & moreover latency period, mode of delivery & preference of care were assessed

ELIGIBILITY:
Inclusion Criteria include women with PPROM ≥28 weeks & <37 weeks with no signs of intra-amniotic infection & membranes rupture is confirmed by a sterile speculum examination and decrease amniotic fluid on ultrasound with singleton, viable, cephalic presenting fetus, morphologically normal fetus by ultrasound & reactive fetal heart rate tracing with no evidence of meconium-stained liquor

Exclusion Criteria:

* Query PPROM: A history of PPROM with no pooling of amniotic fluid from the cervix on a sterile speculum examination
* Maternal comorbidities (Diabetes mellitus, hypertension, etc.)
* Patients with placenta previa
* Amniotic fluid pocket on ultrasound < 2x2 cm
* Logistic problems interfering with follow-up
* Inability to check temperature every six hours, with parameters for notifying their clinician (temperature ≥38°C)
* Non-Dependable transportation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women with rupture of the fetal membranes before 37 weeks of gestation
Study Population: The study will include 3662 women with a history of preterm prelabor rupture of the membranes
Sampling Method: Probability Sample
Enrollment: 3662 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Take-home baby | 2 years
  this outcome is the best indicator of success of the management plan when the outcome is alive & well baby

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine - Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all statistical methods, results of the study ,discussion & recommendations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: onset of January, 2022 (6 months after publication)
Access Criteria: sponsor e.mail & the sponsor organisation
URL: http://www.asu.edu.eg/ar/